CLINICAL TRIAL: NCT07065136
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose and Multiple Ascending Dose Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of SSGJ-627 in Healthy Adult Subjects
Brief Title: Evaluation of 627 in Healthy Adult Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSGJ-627-HV-01
Record Dates: First submitted 2025-04-22; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects (HS)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 627 (Experimental)
  Interventions: Biological: 627; Other: Placebo
- Placebo (Placebo Comparator)
  Interventions: Biological: 627; Other: Placebo

INTERVENTIONS:
Biological: 627 — subcutaneous injection
Other: Placebo — Single subcutaneous injection

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose and multiple ascending dose phase I clinical study to evaluate the safety, tolerability, PK and immunogenicity of SSGJ-627 in healthy adult subjects after single subcutaneous injection.

DETAILED DESCRIPTION:
Seven dose groups are planned for dose escalation in SAD of this study. Subjects in all dose groups will receive a single subcutaneous injection. Group S1 follows open-labeled, single-arm design, Groups S2 to S7 follow randomized, double-blinded, placebo-control design. Blood samples will be collected for PK, immunogenicity, biomarkers, laboratory tests, etc. according to the study schedule throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand protocol requirements and sign a written ICF.
* Male or female subjects aged 18-45 years when signing the ICF.
* Male subjects with body weight ≥ 50 kg, and female subjects with body weight ≥ 45 kg. Subjects with BMI between 18 and 28 kg/m2.
* Subjects whose test results are normal, or abnormal without clinical significance as determined by the investigator.
* Female subjects with childbearing potential and male subjects (and their female partners) must agree to take highly effective contraceptive measures.

Exclusion Criteria:

* History of severe allergy, or with a history of allergy to the study treatment or related excipients.
* History of of significant alcohol abuse.
* History of significant drug abuse.
* Subjects who have positive result for urine nicotine test at screening.
* Pregnant, or nursing females.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | D99
  Incidence of adverse events will be summarized by SOC and PT for each treatment group, and also be summarized by severity and association with the study treatments.